CLINICAL TRIAL: NCT03836482
Title: Feasibility Study to Assess the Safety and Efficacy of a Selective Cytopheretic Device (SCD) to Treat ICU Patients With Acute on Chronic Systolic Heart Failure With Worsening Renal Function Due to Cardiorenal Syndrome or Severe Right Ventricular Failure Awaiting Left Ventricular Assist Device Implantation
Brief Title: Feasibility of the SCD in Cardiorenal Syndrome Patients Awaiting LVAD
Acronym: NEUTRALIZE-CRS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SeaStar Medical (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Michigan (Other); Innovative BioTherapies (IBT) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCD-CRS-01; 1R44HL170779-01A1 (NIH)
Record Dates: First submitted 2019-02-07; First posted 2019-02-11 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-08

CONDITIONS: Acute on Chronic Systolic Congestive Heart Failure; Cardiorenal Syndrome
Keywords: Awaiting Left ventricular assist device implantation; Hospitalized; Selective Cytopheretic Device; SCD; LVAD; CRS
MeSH Terms: conditions — Cardio-Renal Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Selective Cytopheretic Device (Experimental)
  Interventions: Device: Selective Cytopheretic Device

INTERVENTIONS:
Device: Selective Cytopheretic Device — Treatment will be delivered for 4 hours a day for up to 6 consecutive days.

SUMMARY:
Cardiovascular disease is the leading cause of mortality in the US, accounting for 45% of all deaths. Chronic Heart Failure (CHF) is now understood to be a multi-system disease process involving not only the cardiovascular system but also the renal, neuroendocrine, and immune systems. No effective therapy is currently available to treat the most severe subset of CHF patients that have progressed to acute decompensated HF. An innovative approach to reduce the cardio-depressant effects associated with the chronic inflammatory state of CHF may provide a breakthrough for this disorder. This proposal will evaluate the safety and probable benefit to improve cardiac or renal function with an immunomodulatory device to bridge patients to Left Ventricular Assist Device (LVAD) implantation who were previously deemed ineligible for this life sustaining procedure. The Selective Cytopheretic Device (SCD) is an immuno-regulating, extracorporeal membrane device targeted to modulate the cardiodepressant effects assocaited with CHF. SCD is a platform technology focused on immunomodulation of acute and chronic inflammation associated with acute and chronic organ dysfunction. SCD membranes selectively sequester activated systemic leukocytes as they flow through the cartridge via an extracorporeal circuit. Pre-clinical results show that SCD treatment results in a 25% improvement in ejection fraction in a canine CHF model.

This study will enroll 20 patients across up to 5 clinical sites to evaluate the safety and initial efficacy data of SCD treatment in this indication. Patients will receive 4-hour daily SCD treatment for up to 6 days, followed by 6 months of follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 years and older.
2. Evidence of systemic inflammation: blood CRP ≥ 4.5 mg/L or IL-6 ≥ 5.0 pg/ml or neutrophil to lymphocyte ratio ≥3.0.
3. Primary hospitalization for acute decompensated chronic systolic heart failure.
4. Potential LVAD candidate with:

   a) Left ventricular ejection fraction ≤25% (for potential destination therapy) or ≤ 35% (for potential bridge to transplantation) as confirmed by baseline imaging procedure b) NYHA class IIIB or IV chronic (≤ 90 days) systolic heart failure, with failure to respond to optimal medical therapy (beta blocker, ACE inhibitor or ARB or valsartan/sacubitril, aldosterone antagonist, SGLT2i, unless not tolerated or contraindicated, and loop diuretic, as needed) for 45 of the last 60 days c) Known previous peak exercise oxygen consumption < 14 mL/Kg/min or if unable to exercise, dependent on an intra-aortic balloon pump, short-term mechanical circulatory support device or intravenous inotropes unless inotropes contraindicated for clinical reasons (e.g., ventricular arrhythmias)
5. Baseline eGFR** ≥ 40 ml/min/1.73 m2 (baseline defined as the highest known eGFR within 90 days of study enrollment)
6. At least one of the following two criteria:

   1. Severe right ventricular failure (RVF), defined as meeting at least 2 of the following 4 criteria -Central venous pressure > 16 mmHg

      -Central venous pressure/Pulmonary wedge pressure >0.65

      -Right ventricular stroke work index < 300 mmHg * ml/m2

      -Pulmonary artery pulsatility index (PAPi) < 2,
   2. Worsening renal failure (WRF), defined for the purposes of this study as -Increase serum creatinine ≥ 0.5 mg/dL from baseline (baseline defined as the lowest known serum creatinine within 90 days of study enrollment) AND

      * eGFR** ≤ 30 ml/min/1.73 m2 based on serum creatinine at enrollment*** AND
      * Cardiorenal syndrome is the most likely explanation for WRF AND
      * Intolerant or inadequately responsive to standard of care diuretic therapy, defined as persistent signs and/or symptoms of congestion (e.g., peripheral edema, dyspnea, pulmonary rales, neck vein distension) or minimal net volume removal in a 24-hour period despite optimal medical therapy including intravenous diuretic therapy and an estimated need for >5kg fluid removal.

        1. Optimal intravenous diuretic therapy is defined as:

           1. Furosemide equivalent total daily dose of 240mg
           2. Furosemide equivalent dose given either as a single or multiple intravenous bolus or continuous infusion
           3. A furosemide equivalent total daily dose <240mg if the dose has resulted in >3000 mL urine output/24 hours.
7. PA catheter in place at the time of enrollment
8. PCW ≥ 20 mmHg

   * eGFR calculated using the CKD-EPI Creatinine Equation *** Recognizing that this is not a steady state creatinine

Exclusion Criteria:

1. Any clear contraindication to LVAD therapy that is unlikely to resolve with improvement in renal function and volume status
2. Prior sensitivity to dialysis device components
3. Active bacteremia
4. Temperature ≥ 101.5 F or WBC ≥ 10,000 K/uL or any patient with suspected systemic infection.
5. Metastatic malignancy requiring palliative chemo, biologic, or radiation
6. Need for intravenous vasopressor (i.e., phenylephrine, vasopressin), intravenous vasoconstricting inotrope (i.e., norepinephrine or epinephrine) or dopamine > 3 mcg/kg/min. (Note: use of vasodilating inotropes [i.e., dobutamine and milrinone] or dopamine at ≤ 3 mcg/kg/min will not preclude study inclusion)
7. Patients requiring mechanical ventilatory support
8. Patients requiring total parenteral nutrition during the treatment period
9. Persistent SBP < 80 mmHg
10. WBC < 4000 K/uL
11. Platelets < 100,000K/uL
12. Serum creatinine > 4 mg/dL or receiving dialysis / CRRT
13. Acute coronary syndrome within the past month
14. Women who are pregnant, breastfeeding a child, or trying to become pregnant
15. Concurrent enrollment in another interventional clinical trial. Patients enrolled in clinical studies where only measurements and/or samples are taken (i.e., no test device or test drug used) are allowed to participate
16. Use of any other investigational drug or device within the previous 30 days. Patients who participated in a clinical study where only measurements and/or samples are taken (i.e., no test device or drug used) are allowed to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Need for continuous IV vasopressor support | measured daily, at or after 4 hours after termination of daily SCD therapy
  Need for continuous IV vasopressor support with >5 total norepinephrine equivalents and/or >3 vasopressor agents >4 hours following termination of daily SCD therapy session to maintain a MAP >60 mmHg, with norepinephrine equivalents defined as:
  1. 1 x epinephrine (ug/kg/min)
  2. 001 x dopamine (ug/kg/min)
  3. 0.06 x phenylephrine (ug/kg/min)
  4. 2.5 x vasopressin (U/min)
  (Note that use of inotropes (i.e., dobutamine and milrinone) or dopamine at ≤3 mcg/kg/min are not components of this measure.)
Acute myocardial infarction | up to 6 months following SCD treatment initiation
  Acute myocardial infarction as evidenced by elevated cardiac enzymes, with electrocardiographic or imaging findings consistent with myocardial damage and confirmed by Cardiology.
Mortality | up to 6 months following SCD treatment initiation
  Death
Percentage of subjects with reversal of WRF and increase eGFR and PCW | up to 6 days after initiation of SCD therapy
  Among patients with WRF, the percentage of subjects with reversal of WRF (≥ 0.5 mg/dL reduction of serum creatinine from level at study entry), and achieving an eGFR > 30 ml/min/1.73 m2 and PCWP at or below level at study entry at termination of SCD therapy.
Percentage of subjects who no longer have severe right ventricular failure | up to 6 days after initiation of SCD therapy
  Among subjects with severe RVF, the percentage of subjects who no longer have severe right ventricular failure, as evidenced by absence of 3 or more of the following 4 indicators of right ventricular failure:
  1. CVP > 16 mmHg
  2. CVP/PCWP > 0.65
  3. RVSWI < 300 mmHg * mL/m
  4. PAPi < 2
Adverse Events | up to 6 days after initiation of SCD therapy
  Adverse Events due to SCD, hemodialysis catheter, KRT pump, circuit, and hemofilter

SECONDARY OUTCOMES:
Percentage of subject receiving a left ventricular assist device | up to 30 days after the last SCD
Change in 24 hour urine volume | change from onset of intervention to 3 and 6 days after initiation of SCD treatments and from onset of intervention to end of SCD support prior to LVAD implantation
Change in urine sodium | change from onset of intervention to 3 and 6 days after initiation of SCD treatments and from onset of intervention to end of SCD support prior to LVAD implantation
Change in urine creatinine | change from onset of intervention to 3 and 6 days after initiation of SCD treatments and from onset of intervention to end of SCD support prior to LVAD implantation
Change in urine urea | change from onset of intervention to 3 and 6 days after initiation of SCD treatments and from onset of intervention to end of SCD support prior to LVAD implantation
Change in creatinine clearance | change from onset of intervention to 3 and 6 days after initiation of SCD treatments and from onset of intervention to end of SCD support prior to LVAD implantation
Change in urine urea clearance | change from onset of intervention to 3 and 6 days after initiation of SCD treatments and from onset of intervention to end of SCD support prior to LVAD implantation
Change in Pulmonary Capillary Wedge Pressure (PCWP) | change from onset of intervention to 3 and 6 days after initiation of SCD treatments and from onset of intervention to end of SCD support prior to LVAD implantation
  If PCWP cannot be obtained, Pulmonary Artery Diastolic Pressure (PADP) will be used in its place. When utilizing PADP in place of PCWP for change measures, comparisons will be made to baseline PADP.
Change in serum sodium | change from onset of intervention to 3 and 6 days after initiation of SCD treatments and from onset of intervention to end of SCD support prior to LVAD implantation
Change in serum potassium | change from onset of intervention to 3 and 6 days after initiation of SCD treatments and from onset of intervention to end of SCD support prior to LVAD implantation
Change in serum dissolved carbon dioxide (CO2) | change from onset of intervention to 3 and 6 days after initiation of SCD treatments and from onset of intervention to end of SCD support prior to LVAD implantation
Change in blood urea nitrogen (BUN) | change from onset of intervention to 3 and 6 days after initiation of SCD treatments and from onset of intervention to end of SCD support prior to LVAD implantation
Change in serum creatinine | change from onset of intervention to 3 and 6 days after initiation of SCD treatments and from onset of intervention to end of SCD support prior to LVAD implantation
Percentage of subjects with reduction of serum creatinine (≥ 0.5 mg/dL) and PCWP (≤ 18 mmHg) | change from onset of intervention to 3 and 6 days after initiation of SCD treatments and from onset of intervention to end of SCD support prior to LVAD implantation
  If PCWP cannot be obtained, PADP will be used in its place. When utilizing PADP in place of PCWP for change measures, comparisons will be made to baseline PADP
Percentage of subjects receiving a left ventricular assist device with serum creatinine ≥ 0.5 mg/dL below level at study entry | 30 days following discontinuation of SCD
Change in right ventricular fractional area change | change from onset of intervention to 3 and 6 days after initiation of SCD treatments and from onset of intervention to end of SCD support prior to LVAD implantation
  Change in right ventricular fractional area change, TAPSE, and right ventricular global longitudinal strain

IPD SHARING:
Plan to Share IPD: Undecided